CLINICAL TRIAL: NCT05895669
Title: Evaluation of Cardiovascular Outcomes in Patients Undergoing Orthotopic Liver Transplantation: a Retrospective Cohort Study
Brief Title: Cardiovascular Outcomes in Orthotopic Liver Transplanted Patients (COLT Study)
Acronym: COLT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Alfredo Caturano, Principal Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: 0012771/i
Record Dates: First submitted 2023-05-26; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Liver Transplant; Complications; Cardiovascular Complication; Cardiovascular; Attack; Cardiovascular Stroke; Death
MeSH Terms: conditions — Myocardial Infarction; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All patients with orthotopic liver transplantation who are evaluated and followed at each participating centers will be recorded in this study. Within this register a characterization of patients and therapy will be done. Prognostic factors of defined clinical relevant endpoints will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All patients with ortothopic liver transplantation and at least 2 year follow-up at the referral center

Exclusion Criteria:

* Missing Informed Consent Form
* Missing Contact Informations for Follow up

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with ortothopic liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-05-02 (Estimated); Study Completion 2024-05-02 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular death | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  death due to cardiac causes (myocardial infraction and/or stroke)
cardiovascular complication | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  fatal and non fatal myocardial infraction and/or stroke

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Gragnano Hospital, Gragnano, SA
  - University of Campania Luigi Vanvitelli, Napoli

IPD SHARING:
Plan to Share IPD: Undecided